CLINICAL TRIAL: NCT06209255
Title: Case Report: Treatment of Hip Instability After Total Hip Replacement With Pelvic Osteotomy Using A Modified Stoppa Approach
Brief Title: Pelvic Osteotomy Of The Total Hip Replacement
Status: Completed | Type: Observational
Sponsor: Van Bölge Eğitim ve Araştırma Hastanesi (Other Government)
Responsible Party: Principal Investigator, Javad Mirzazada, MD, Orthopedics And Traumathology Specialist, Van Bölge Eğitim ve Araştırma Hastanesi
Other Study IDs: VanBEAH
Record Dates: First submitted 2023-12-04; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Congenital Hip Dysplasia; Hip Osteoarthritis
Keywords: revision hip arthroplasty
MeSH Terms: conditions — Hip Dislocation, Congenital; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pelvic Osteotomy - Ganz Procedure — Ischial osteotomy was performed on the pubic arch; this was followed by iliac osteotomy, performed using Schanz screws in the iliac wing. The osteotomized acetabulum was overturned, and inclination was reduced.

SUMMARY:
This observational study aims to learn about the outcomes in the previously operated patient and whether pelvic bone rearrangement surgery was a success.

The main question it aims to answer is:

• Should the investigators perform pelvic rearrangement surgery on a patient if there's not enough bone stock to accomplish the exchange of the components?

As the research started the participant was asked to attend outpatient clinics regularly and keep in touch. The investigators were able to observe the outcomes and closely explore probable risks for failure.

DETAILED DESCRIPTION:
A 56-year-old female patient had a hip operation one year previously and experienced her first dislocation two months postoperatively. The patient underwent closed reduction three times. The patient presented to us due to a fourth hip dislocation that had occurred one month previously. Hip X-ray images revealed acetabular component malposition, with an 80-degree inclination and 20 degrees of cup anteversion with a posterior hip dislocation. The investigators treated the patient via pelvic osteotomy, using a modified Stoppa approach to reduce acetabular inclination. The patient had no dislocation at the 2-year follow-up. At the last follow-up, the Harris Hip Score was 85.

ELIGIBILITY:
Inclusion Criteria:

* Previously Replaced Total Hip
* Minimum 1-year follow-up
* 18-45 years, both sexes
* otherwise healthy

Exclusion Criteria:

* Any debilitating disorder
* Neurological or genetic disorders
* Pediatric or geriatric age

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Since this is a single-case observational study, a population description could not be made.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | 3 years
  Higher scores, the better.

SECONDARY OUTCOMES:
Visual Analogue Score | 3 years
  Lower the scores, the better.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Coskun, MD, Principal Investigator — Physician
Locations (1):
- VanBEAH, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kocabiyik A, Misir A, Kizkapan TB, Yildiz KI, Kaygusuz MA, Alpay Y, Ezici A. Changes in Hip, Knee, and Ankle Coronal Alignments After Total Hip Arthroplasty With Transverse Femoral Shortening Osteotomy for Unilateral Crowe Type IV Developmental Dysplasia of the Hip. J Arthroplasty. 2017 Nov;32(11):3449-3456. doi: 10.1016/j.arth.2017.05.044. Epub 2017 Jun 1. PMID 28641973
- [Background] Guo L, Yang Y, An B, Yang Y, Shi L, Han X, Gao S. Risk factors for dislocation after revision total hip arthroplasty: A systematic review and meta-analysis. Int J Surg. 2017 Feb;38:123-129. doi: 10.1016/j.ijsu.2016.12.122. Epub 2016 Dec 31. PMID 28043927
- [Background] Yetkin C, Yildirim T, Alpay Y, Tas SK, Buyukkuscu MO, Dirvar F. Evaluation of Dislocation Risk Factors With Total Hip Arthroplasty in Developmental Hip Dysplasia Patients: A Multivariate Analysis. J Arthroplasty. 2021 Feb;36(2):636-640. doi: 10.1016/j.arth.2020.08.043. Epub 2020 Aug 29. PMID 32943316
- [Background] Alberton GM, High WA, Morrey BF. Dislocation after revision total hip arthroplasty : an analysis of risk factors and treatment options. J Bone Joint Surg Am. 2002 Oct;84(10):1788-92. PMID 12377909
- [Background] Sadhu A, Nam D, Coobs BR, Barrack TN, Nunley RM, Barrack RL. Acetabular Component Position and the Risk of Dislocation Following Primary and Revision Total Hip Arthroplasty: A Matched Cohort Analysis. J Arthroplasty. 2017 Mar;32(3):987-991. doi: 10.1016/j.arth.2016.08.008. Epub 2016 Aug 20. PMID 27633947
- [Background] Ballester Alfaro JJ, Sueiro Fernandez J. Trabecular Metal buttress augment and the Trabecular Metal cup-cage construct in revision hip arthroplasty for severe acetabular bone loss and pelvic discontinuity. Hip Int. 2010;20 Suppl 7:S119-27. doi: 10.1177/11207000100200s720. Epub 2010 May 27. PMID 20512783
- [Background] Dennis DA. Management of massive acetabular defects in revision total hip arthroplasty. J Arthroplasty. 2003 Apr;18(3 Suppl 1):121-5. doi: 10.1054/arth.2003.50105. PMID 12730946
- [Background] DeBoer DK, Christie MJ, Brinson MF, Morrison JC. Revision total hip arthroplasty for pelvic discontinuity. J Bone Joint Surg Am. 2007 Apr;89(4):835-40. doi: 10.2106/JBJS.F.00313. PMID 17403808
- [Background] Sheth NP, Nelson CL, Springer BD, Fehring TK, Paprosky WG. Acetabular bone loss in revision total hip arthroplasty: evaluation and management. J Am Acad Orthop Surg. 2013 Mar;21(3):128-39. doi: 10.5435/JAAOS-21-03-128. PMID 23457063
- [Background] Paprosky WG, Perona PG, Lawrence JM. Acetabular defect classification and surgical reconstruction in revision arthroplasty. A 6-year follow-up evaluation. J Arthroplasty. 1994 Feb;9(1):33-44. doi: 10.1016/0883-5403(94)90135-x. PMID 8163974
- [Background] Malahias MA, Ma QL, Gu A, Ward SE, Alexiades MM, Sculco PK. Outcomes of Acetabular Reconstructions for the Management of Chronic Pelvic Discontinuity: A Systematic Review. J Arthroplasty. 2020 Apr;35(4):1145-1153.e2. doi: 10.1016/j.arth.2019.10.057. Epub 2019 Nov 4. PMID 31784362